CLINICAL TRIAL: NCT00524563
Title: Clinical Outcomes and Global Epidemiology -Data Coordinating Center
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Sponsor
Other Study IDs: PRO07080042
Record Dates: First submitted 2007-08-31; First posted 2007-09-03 (Estimated); Last update posted 2018-06-12 (Actual); Status verified 2018-06

CONDITIONS: Acinetobacter Infections
Keywords: Acinetobacter; bloodstream infection; Isolate
MeSH Terms: conditions — Acinetobacter Infections; Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The primary objective is to assess for independent predictors of in-hospital mortality (up to 28 days) in patients with Acinetobacter bloodstream infection. Secondary Objectives include the following: To determine the impact of inactive empiric antimicrobial therapy, defined as receipt of empiric antimicrobial therapy with no in vitro activity against the offending isolate for at least 24hrs, on the outcome (end points defined below) of patients with Acinetobacter bloodstream infection. To determine the impact of carbapenem resistance and pan-drug resistance (defined as resistance to all antimicrobials except colistin and/or tigecycline if these agents were tested) on the outcome of patients with Acinetobacter bloodstream infection. To assess the efficacy of varying definitive therapies on the outcome of patients with Acinetobacter bloodstream infection. To characterize the molecular epidemiology of Acinetobacter on a global level, as determined by pulsed-field gel electrophoresis (PFGE) and other techniques, and to assess whether patient outcomes are clonally related and to characterize the mechanisms of resistance in Acinetobacter on a global scale.

DETAILED DESCRIPTION:
Medical records will be reviewed and information collected from charts to assess for independent predictors of in-hospital mortality (up to 28 days) in patients with Acinetobacter bloodstream infection. 24 sites will participate and all information will be loaded into a password protected database.

ELIGIBILITY:
Inclusion Criteria:

* Acinetobacter bloodstream infection

Exclusion Criteria:

* Does not meet entry criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: acinetobacter infection
Sampling Method: Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2007-07 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Paterson, MD, Principal Investigator — University of Pittsburgh Medical Center
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States